CLINICAL TRIAL: NCT00991263
Title: Intrinsic Breast Cancer Subtypes and Benefit of Paclitaxel in CALGB 9344 and Dose Dense Therapy in CALGB 9741
Brief Title: Study of Tissue Samples From Women Treated With Paclitaxel for Breast Cancer on Clinical Trial CALGB-9344 or CALGB-9741
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-159905C-ICSC; CALGB-159905C-ICSC; CDR0000647570 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Tissue blocks from CALGB-9344 and CALGB-9741 are utilized to purify RNA to be tested in the PAM50 assay (a 50-gene quantitative PCR assay, that provides an intrinsic breast cancer subtype diagnosis) and generate risk of relapse (ROR) scores. For more information, see Details section.
  Interventions: Genetic: gene expression analysis; Genetic: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at tissue samples from women treated with paclitaxel for breast cancer on clinical trial CALGB 9344 or CALGB 9741.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether subtype-specific treatment effects correlate with disease-free survival (DFS), as determined by a significant interaction between PAM50-based intrinsic subtypes, and (a) paclitaxel benefit in CLB-9344 and (b) dose density in CALGB-9741.
* To determine whether subtype-specific treatment effects correlate with DFS for the HER2-negative subsets in CALGB-9344 and CALGB-9741, as determined by analysis of tissue microarray (TMA) and slides.
* To determine the relationship between PAM50-defined risk of relapse (ROR) score and DFS in CALGB-9344 and CALGB-9741.
* To evaluate the relationship between PAM50-defined ROR score and DFS in the HER2-negative subsets in CALGB-9344 and CALGB-9741, as determined by analysis of TMA and slides.
* To examine the relationship between PAM50-defined proliferation score and DFS in CALGB-9344 and CALGB-9741 in multivariate Cox-proportional hazards models including the following covariates: (a) number of positive lymph nodes, square root transformation; (b) menopausal status (pre versus peri/post); CALGB-9344 only; c) dose of doxorubicin hydrochloride (60/75/90 mg/m^2); and CALGB-9741 only; and (d) sequence of treatment.

Secondary

* To evaluate overall survival (OS) in a Cox-proportional hazards-regression model for testing the interaction between ROR with (a) paclitaxel benefit in CALGB-9344 and (b) dose density in CALGB-9741.
* To test for a significant interaction between ROR and paclitaxel benefit at 5-year and 10-year DFS.
* To test whether 5-year and 10-year DFS rates can be associated to a significant interaction between the proliferation score with (a) paclitaxel benefit in CALGB-9344 and (b) dose density in CALGB-9741.

OUTLINE: Tissue blocks from CALGB-9344 and CALGB-9741 are utilized to purify RNA to be tested in the PAM50 assay (a 50-gene quantitative PCR assay, that provides an intrinsic breast cancer subtype diagnosis) and generate risk of relapse (ROR) scores.

The assay identifies five subtypes with the following characteristics:

* Luminal A: This subtype expresses estrogen receptor (ER) accompanied by high levels of ER-associated gene expression. Genes associated with cell cycle activation are not highly expressed and this tumor type is only very rarely HER2+. This subgroup has the most favorable prognosis and is enriched for endocrine therapy responsive tumors.
* Luminal B: This subtype expresses ER and ER-associated gene expression but to a lower extent. Genes associated with cell cycle activation are highly expressed and this tumor type can be HER2+ (~20%) or HER2- thus, from the clinical perspective, Luminal B tumors are at least two further subtypes defined by the presence or absence of HER2-gene amplification. The prognosis is unfavorable (despite ER expression) and endocrine therapy responsiveness is generally diminished.
* Basal-like: This subtype is ER-, is almost always clinically HER2- and expresses a suite of "basal" biomarkers. Genes associated with cell cycle activation are highly expressed.
* HER2-enriched: This subtype is ER- and is HER2+ in the majority of cases. Genes associated with cell cycle activation are highly expressed and these tumors have a poor outcome. Tumors within this classification that are clinically HER2- fall into a class previously described as double-negative non-basal.
* Normal-like: A tumor subtype diagnosis cannot be provided from samples that exhibit a normal-like profile. Since this profile was trained on samples without cancer, "normal-like" implies there are too few tumor cells in the sample to make a true tumor subtype diagnosis.

PROJECTED ACCRUAL: A total of 2,245 tissue blocks from CALGB-9544 and 1,432 tissue blocks from CALGB-9741 will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage II or IIIA breast cancer

  * Received treatment with paclitaxel on clinical trial CALGB-9344 or CALGB-9741
* Tissue blocks available

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Pre-, peri-, or postmenopausal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer previously treated with paclitaxel and enrolled on CALGB-9344 or CALGB-9741.
Sampling Method: Non-Probability Sample
Enrollment: 3677 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 10 years

SECONDARY OUTCOMES:
5- and 10-year DFS rates | Up to 10 years
Overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Ellis, MD, PhD, FRCP, Study Chair — Washington University Siteman Cancer Center